CLINICAL TRIAL: NCT06825208
Title: Etoposide Plus Benmelstobart Followed by Maintenance Therapy of Benmelstobart Plus Anlotinib in First-line Treatment of Elderly Patients with Extensive Stage Small Cell Lung Cancer: a Single-arm, Prospective Trial
Status: Not yet recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Fangsurong, Head of the Department of Respiratory and Critical Care Medicine, Nanjing First Hospital, Nanjing Medical University
Other Study IDs: 2450-E-A-ES-SCLC-001
Record Dates: First submitted 2025-02-09; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Small Cell Lung Cancer Extensive Stage; ELDERLY PEOPLE

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Elderly patients with extensive stage small cell lung cancer: Elderly patients with extensive small-cell lung cancer who have not previously received systematic treatment

SUMMARY:
This is a prospective, single-arm clinical study to evaluate the efficacy and safety of etoposide in combination with bemosubezumab and sequential Benmelstobart in combination with Anlotinib as first-line treatment for elderly patients with extensive small-cell lung cancer.

Participants who met the inclusion criteria were selected to enter the study and received etoposide combined with Benmelstobart followed by bemosubezumab combined with Anlotinib. The primary endpoint was PFS (Progression-free Survival), the secondary endpoint was OS (Overall Survival) and safety (CTCAE 5.0), and the exploratory endpoint was the screening of various potential molecular markers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathologically proven extensive small-cell Lung cancer (according to the Veterans Administration Lung Study Group, VALG stage) who have not previously received systematic treatment for extensive small-cell lung cancer;
* Patients who have previously received chemoradiotherapy for limited-stage SCLC must have received radical therapy and have at least 6 months of treatment-free intervals between the end of chemotherapy, radiotherapy, or chemoradiotherapy and the diagnosis of extensive SCLC (end time of last chemotherapy cycle/end time of last radiotherapy).
* There was no gender limitation. The subjects voluntarily joined the study, signed the informed consent, and the compliance was good
* Aged eligibility criteria are considered to be met if the following criteria are met:

Patient requirements: Between 70 and 85 years old, and after independent assessment by two chief physicians, the patient's physical condition may not be able to tolerate platinum-containing chemotherapy regimen, and the patient's informed consent to accept the platinum treatment regimen;

* ECOG score: 0-2;
* At least one lesion can be measured by CT.
* Expect to survive for at least 3 months.
* The main organ functions within 7 days before treatment should meet the following criteria:

  1) Blood routine examination (under the condition of no blood transfusion or use of hematopoietic stimulating factor drugs for correction within 14 days): Hemoglobin (Hb) ≥ 90g/L; Absolute neutrophil count (ANC) ≥ 1.5×109/L; ； 1) Platelet count (PLT) ≥ 100×10⁹/L; white blood cell count (WBC) ≥ 3.0×10⁹/L.

  2) Biochemical tests: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN (for patients with liver metastasis from tumors, ≤ 5×ULN); total bilirubin (TBIL) ≤ 1.5×ULN (for Gilbert's syndrome patients, ≤ 3×ULN); serum creatinine (Cr) ≤ 1.5×ULN or creatinine clearance rate ≥ 50 ml/min; 3) Coagulation function: activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT) ≤ 1.5×ULN; 4) Doppler ultrasound assessment: Left ventricular ejection fraction (LVEF) ≥ 50%. 。
* Men should agree that contraception must be used during the study period and for 6 months after the end of the study period;

Exclusion Criteria:

* Used antiangiogenic drugs or related immunotherapy drugs such as PD-1 and PD-L1 in the past;
* Subjects with known central nervous system metastatic and/or cancerous meningitis; (Unless asymptomatic, or treated and stable, no radiographic evidence of new BMS or enlarged BMS was found at least 2 weeks after BMS treatment, and steroid or anticonvulsant therapy was discontinued for at least 14 days before study therapy began. If active or new untreated, asymptomatic CNS metastases are found on imaging in subjects during the screening period, radiation therapy or untreated imaging evidence of new or enlarged BMS is required for at least 2 weeks.)
* Subject has had or co-developed other malignancies (except cured basal cell carcinoma of the skin and cervical carcinoma in situ) within 5 years;
* Subject has multiple factors that affect oral medication (such as inability to swallow, post-gastrointestinal resection, chronic diarrhea, and intestinal obstruction);
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
* Spinal cord compression that has not been cured or alleviated by surgery and/or radiotherapy, or previously diagnosed spinal cord compression with no clinical evidence of disease stabilization ≥1 week prior to randomization after treatment;
* Imaging (CT or MRI) shows that the tumor invades the large blood vessels or has an unclear boundary with the large blood vessels;
* Subjects with evidence or history of bleeding tendencies, regardless of severity, within 2 months prior to initial dosing; A history of hemoptysis (defined as bright red or 1/2 teaspoon of blood) or unhealed wounds, ulcers, or fractures within 2 weeks prior to initial medication;
* Subjects whose adverse events (other than alopecia) from prior treatment did not recover to ≤CTCAE Class 1;
* Received major surgical treatment or significant traumatic injury within 28 days prior to randomization;
* Those who had experienced an arterial/venous thrombosis event, such as cerebrovascular accident (including temporary ischemic attack), deep vein thrombosis and pulmonary embolism, within 6 months before randomization;
* have a history of psychotropic drug abuse and can not quit or have mental disorders;
* Subjects with any severe and/or uncontrolled medical condition, including:

  a) Subjects with unsatisfactory blood pressure control (systolic ≥150 mmHg or diastolic ≥100mmHg); b) have grade 2 myocardial ischemia or myocardial infarction, arrhythmias (including QTc≥450ms in men, QTc≥ 470ms in women), and grade 2 congestive heart failure (NYHA); c) Active or uncontrolled severe infection (≥CTC AE grade 2 infection); d) Cirrhosis, active hepatitis *;

  * Active hepatitis (Hepatitis B reference :HBsAg positive, and HBV DNA test value exceeds the upper limit of normal; Hepatitis C reference :HCV antibody positive, and HCV virus titer test value exceeds the upper limit of normal value); e) HIV positive test; f) Poor diabetes control (fasting blood glucose (FBG)>10mmol/L); g) Urine routine indicated urine protein ≥++, and confirmed 24-hour urine protein quantity >1.0 g;
* have received prophylactic or attenuated vaccine within 4 weeks before the first dose;
* Severe hypersensitivity after administration of other monoclonal antibodies;
* The need for systemic treatment (e.g., use of disease-modifying drugs, Active autoimmune diseases with corticosteroids or immunosuppressants (e.g., but not limited to: autoimmune hepatitis, interstitial pneumonia, enteritis, vasculitis, nephritis; Patients with asthma requiring medical intervention with bronchodilators were not included). Replacement therapies (such as thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) are not considered systemic.
* have been diagnosed with an immune deficiency or are receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy (dose >10mg/ day prednisone or other therapeutic hormone) and continue to use within 2 weeks before the first dose;
* Have participated in other clinical trials within four weeks;
* concomitant diseases that, in the investigator's judgment, seriously endanger the safety of the subject or interfere with the patient's completion of the study.

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients from Nanjing First Hospital
Sampling Method: Non-Probability Sample
Enrollment: 29 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival time | From enrollment to the end of treatment at 18 months
  It is the time that passes from a certain date (generally the first day of treatment, or the day in which a patient is enrolled in a clinical trial) and the date on which disease "progresses" or the date on which the patient dies, from any cause.

IPD SHARING:
Plan to Share IPD: No